CLINICAL TRIAL: NCT02184988
Title: A Multi-center, Open Label, Multiple Dose, Phase II Trial to Demonstrate the Safety of DWP-450 in Adult Subjects for Treatment of Moderate-to-severe Glabellar Lines.
Brief Title: Safety Study of DWP-450 (Botulinum Purified Neurotoxin, Type A) Injection to Treat Glabellar Lines
Acronym: EV-004
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Evolus, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Evolus - CLIN004
Record Dates: First submitted 2014-07-02; First posted 2014-07-09 (Estimated); Results first posted 2019-02-05 (Actual); Last update posted 2019-04-24 (Actual); Status verified 2019-04

CONDITIONS: Glabellar Frown Lines
Keywords: Glabellar Lines; Botulinum purifies neurotoxin, Type A (DWP-450)
MeSH Terms: interventions — DWP450; Injections

STUDY DESIGN:
Masking Description: Open Label
Oversight: Data Monitoring Committee: No

ARMS (1):
- Botulinum neurotoxin, Type A (Experimental): DWP-450 (Botulinum purified neurotoxin, Type A) Injection
  Interventions: Biological: Botulinum purified neurotoxin, Type A

INTERVENTIONS:
Biological: Botulinum purified neurotoxin, Type A — The subject is to be injected intra-muscularly into a total of five sites: the mid-line of the procures muscle, the inferomedial aspect of each corrugator muscle and the superior middle aspect of each corrugator, at least 1 cm above the bony orbital rim. Each site is injected with 0.1 ml (4U), for a total of 20 U and 0.5 ml.
  Other Names: DWP-450 (Botulinum purified neurotoxin, Type A) Injection

SUMMARY:
The purpose of this study is to demonstrate the safety of multiple doses of DWP-450 (Botulinum purified neurotoxin, Type A) Injection in treatment of moderate to severe glabellar lines in adult subjects.

DETAILED DESCRIPTION:
Three hundred and fifty subjects will be enrolled and injected with the study drug DWP-450 over the course of the 365 day study.

Subjects with moderate or severe glabellar lines at maximum frown on the 4 point Glabellar Line Scale (GLS, 0=none, 1= mild, 2=moderate, 3=severe), as judged by the investigator, will be eligible for injection with DWP-450. After each injection, subjects will be followed and are eligible for a repeat injection if their GLS is ≥2 at maximum frown, as judged by the Investigator. If a subject does not have a GLS≥2 they will be followed monthly until eligible for repeat treatment.

Subjects may receive up to a maximum of 4 treatments and will be followed for 365 days from initial treatment.

ELIGIBILITY:
Inclusion Criteria (A subject must meet all of the following inclusion criteria in order to be eligible for enrollment in the study):

* Subjects must be an adult 18 years of age or over
* Subject is able to provide informed consent and comply with study instructions
* Subject has moderate to severe glabellar lines on maximum frown as assessed by the investigator using the GLS
* Subject is willing and able to complete the entire course of the study

Exclusion Criteria (A subject must not meet the following exclusion criteria in order to be eligible for enrollment in the stud)y:

* Previous treatment with botulinum toxin of any serotype in the forehead area within the last 8 months
* Previous treatment with any facial aesthetic procedure (e.g. injection with fillers, chemical peeling, photo rejuvenation) in the glabellar area within the last 12 months
* Previous insertion of permanent material in the glabellar area
* Planned treatment with botulinum toxin of any serotype in any other body region during the study period
* Any surgery in the glabellar area including surgical removal of the corrugator, procerus, or depressor supercilii muscles or a combination of these, or scars in the glabellar area and the surrounding areas (including eye brow)
* Energy based or cryo-therapy based treatment of facial muscles superior to the lateral canthus
* Any other planned facial aesthetic procedure during the trial period, superior to the level of the lateral canthus (subjects can continue with their usual skin care routine)
* Inability to substantially lessen glabellar frown lines even by physically spreading them apart
* Marked facial asymmetry
* Ptosis of eyelid and/or eyebrow, or history of eyelid and/or eyebrow ptosis
* History of facial nerve palsy
* Excessive dermatochalasis, deep dermal scarring, thick sebaceous skin
* Any active infection in the area of the injection sites
* Medical condition that may affect neuromuscular function (e.g., myasthenia gravis, Eaton-Lambert syndrome, amyotrophic lateral sclerosis)
* Evidence of recent alcohol or drug abuse
* Medical or psychiatric conditions that may increase the risk associated with study participation or may interfere with the interpretation of study results and, in the judgment of the Investigator, would make the subject inappropriate for entry into this study
* Pregnant or sexually active female subjects who are of childbearing potential and who are not willing to use an acceptable form of contraception
* Known allergy or hypersensitivity to botulinum toxin preparation
* Participation in another interventional clinical study within the last 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 352 (Actual)
Dates: Start 2014-08; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rui Avelar, MD, Study Director — Evolus, Inc.
Locations (1):
- ATS Clinical Research, Santa Monica, California, United States

IPD SHARING:
Plan to Share IPD: No
Analysis will be of combined data for all subjects entered into the study

REFERENCES:
- [Derived] Nam HS, Park YG, Paik NJ, Oh BM, Chun MH, Yang HE, Kim DH, Yi Y, Seo HG, Kim KD, Chang MC, Ryu JH, Lee SU. Efficacy and safety of NABOTA in post-stroke upper limb spasticity: a phase 3 multicenter, double-blinded, randomized controlled trial. J Neurol Sci. 2015 Oct 15;357(1-2):192-7. doi: 10.1016/j.jns.2015.07.028. Epub 2015 Jul 21. PMID 26233808

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Botulinum Neurotoxin, Type A
Started | 352
Completed | 297
Not Completed | 55
Not completed — Pregnancy | 2
Not completed — Adverse Event | 2
Not completed — moving away/travelling/unable to complet | 6
Not completed — work scheduling issues | 4
Not completed — various other reasons | 9
Not completed — Lost to Follow-up | 32

BASELINE CHARACTERISTICS:
Arm/Group | Botulinum Neurotoxin, Type A
Number analyzed (Participants) | 352
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 319
  >=65 years | 33
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 331
  Male | 21

OUTCOME MEASURES:

1. Primary Outcome: The Safety of Repeat DWP-450 Treatments - Proportion of Subjects With at Least One Adverse Event Over 1 Year
Description: The primary safety analysis was the calculation of the proportion of subjects with at least one adverse event that occurred from Day 0 through Day 365.
Time Frame: 365 Days
Measure: Count of Participants; unit: Participants
Arm/Group | Botulinum Neurotoxin, Type A
Number analyzed (Participants) | 352
Participants | 148

2. Other Pre Specified Outcome: Percentage of Subjects With an Improvement of 1 Point or More (i.e., ≥1 Point Responders) at Rest on Day 365, by Investigator Assessment on the Glabellar Line Scale (GLS)
Description: GLS is scored: 0=none, 1=mild, 2=moderate, 3=severe. A 1-point decrease in GLS score is equivalent to a 1-point improvement on the GLS; as such, both meet the definition of a 1-point responder on the GLS
Time Frame: 365 Days
Population: 323 subjects had a GLS score at rest >0 (i.e., 1, 2 or 3) at baseline and therefore could potentially have had a ≥1 point improvement in GLS score at rest at a post-baseline visit; 32 were missing the EOS GLS assessment
Measure: Number (95% Confidence Interval); unit: percentage of responders
Arm/Group | Botulinum Neurotoxin, Type A
Number analyzed (Participants) | 291
percentage of responders | 75.9 [70.6 to 80.7]

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Botulinum Neurotoxin, Type A
All-Cause Mortality (participants affected / at risk) | 0/352
Serious Adverse Events (participants affected / at risk) | 7/352
Other Adverse Events (participants affected / at risk) | 141/352
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Botulinum Neurotoxin, Type A (N=352)
Device failure - failure of pacemaker/defibrillator (General disorders) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Malignant anorectal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Dysfunctional uterine bleeding (Reproductive system and breast disorders) | 1 (2)
Ovarian Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Botulinum Neurotoxin, Type A (N=352)
Headache (Nervous system disorders) | 54 (65)
Lethargy (Nervous system disorders) | 2 (2)
Muscle tone disorder (Nervous system disorders) | 2 (2)
Sinus headache (Nervous system disorders) | 2 (2)
Speech disorder (Nervous system disorders) | 2 (2)
Dizziness (Nervous system disorders) | 1 (1)
Migraine (Nervous system disorders) | 1 (1)
Migraine with aura (Nervous system disorders) | 1 (1)
Nerve compression (Nervous system disorders) | 1 (1)
Paresthesia (Nervous system disorders) | 1 (1)
Post herpetic neuralgia (Nervous system disorders) | 1 (1)
Thoracic outlet syndrome (Nervous system disorders) | 1 (1)
Bronchitis (Infections and infestations) | 8 (8)
Diverticulitis (Infections and infestations) | 2 (2)
Influenza (Infections and infestations) | 9 (9)
Gastroenteritis viral (Infections and infestations) | 5 (5)
Nasopharyngitis (Infections and infestations) | 4 (4)
Sinusitis (Infections and infestations) | 12 (12)
Tooth infection (Infections and infestations) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 4 (4)
Urinary tract infection (Infections and infestations) | 9 (9)
abscess limb (Infections and infestations) | 1 (1)
cystitis (Infections and infestations) | 1 (1)
ear infection (Infections and infestations) | 1 (1)
herpes zoster (Infections and infestations) | 1 (1)
laryngitis (Infections and infestations) | 1 (1)
oral candidiasis (Infections and infestations) | 1 (1)
oral herpes (Infections and infestations) | 1 (1)
pharyngitis (Infections and infestations) | 1 (1)
pharyngitis streptococcal (Infections and infestations) | 1 (1)
tinea faciei (Infections and infestations) | 1 (1)
viral infection (Infections and infestations) | 1 (1)
Influenza like illness (General disorders) | 2 (2)
Injection site bruising (General disorders) | 4 (4)
Injection site pain (General disorders) | 4 (4)
chest pain (General disorders) | 1 (1)
fatigue (General disorders) | 1 (1)
injection site cyst (General disorders) | 1 (1)
injection site laceration (General disorders) | 1 (1)
injury associated with a device (General disorders) | 1 (1)
Asthenopia (Eye disorders) | 2 (3)
Blepharospasm (Eye disorders) | 1 (1)
Dry eye (Eye disorders) | 1 (1)
Eyelid edema (Eye disorders) | 2 (2)
Eyelid ptosis (Eye disorders) | 5 (5)
Lacrimation increased (Eye disorders) | 2 (2)
Presbyopia (Eye disorders) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (2)
arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
bursitis (Musculoskeletal and connective tissue disorders) | 1 (1)
myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1)
pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
pain in jaw (Musculoskeletal and connective tissue disorders) | 1 (1)
rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1)
tenosynovitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 2 (2)
Meniscus injury (Injury, poisoning and procedural complications) | 2 (2)
arthropod bite (Injury, poisoning and procedural complications) | 1 (1)
fall (Injury, poisoning and procedural complications) | 1 (1)
incision site pain (Injury, poisoning and procedural complications) | 1 (1)
limb injury (Injury, poisoning and procedural complications) | 1 (1)
lip injury (Injury, poisoning and procedural complications) | 1 (1)
median nerve injury (Injury, poisoning and procedural complications) | 1 (1)
post procedural swelling (Injury, poisoning and procedural complications) | 1 (1)
road traffic accident (Injury, poisoning and procedural complications) | 1 (1)
thermal burn (Injury, poisoning and procedural complications) | 1 (1)
wrist fracture (Injury, poisoning and procedural complications) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 2 (2)
diarrhea (Gastrointestinal disorders) | 1 (1)
dyspepsia (Gastrointestinal disorders) | 1 (1)
gastro-esophageal reflux disease (Gastrointestinal disorders) | 1 (1)
large intestine polyp (Gastrointestinal disorders) | 1 (1)
nausea (Gastrointestinal disorders) | 1 (1)
pancreatic cyst (Gastrointestinal disorders) | 1 (1)
pancreatic pseudocyst (Gastrointestinal disorders) | 1 (1)
toothache (Gastrointestinal disorders) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Melanocytic nevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
benign breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 (2)
acne (Skin and subcutaneous tissue disorders) | 1 (1)
dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1)
ecchymosis (Skin and subcutaneous tissue disorders) | 1 (1)
psoriasis (Skin and subcutaneous tissue disorders) | 1 (1)
rosacea (Skin and subcutaneous tissue disorders) | 1 (1)
skin tightening (Skin and subcutaneous tissue disorders) | 1 (1)
skin wrinkling (Skin and subcutaneous tissue disorders) | 1 (1)
Depression (Psychiatric disorders) | 2 (2)
Insomnia (Psychiatric disorders) | 2 (2)
anxiety (Psychiatric disorders) | 1 (1)
ADHD (Psychiatric disorders) | 1 (1)
decreased appetite (Metabolism and nutrition disorders) | 1 (1)
diabetes mellitus (Metabolism and nutrition disorders) | 1 (1)
hypercholesterolemia (Metabolism and nutrition disorders) | 1 (1)
hyperlipidemia (Metabolism and nutrition disorders) | 1 (1)
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1)
cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
vulvovaginal swelling (Reproductive system and breast disorders) | 1 (1)
hypertension (Vascular disorders) | 4 (4)
atrial tachycardia (Cardiac disorders) | 1 (1)
palpitations (Cardiac disorders) | 1 (1)
hypersensitivity (Immune system disorders) | 1 (1)
seasonal allergy (Immune system disorders) | 1 (1)
ear congestion (Ear and labyrinth disorders) | 1 (1)
glucose in urine (Investigations) | 1 (1)
nephrolithiasis (Renal and urinary disorders) | 2 (2)
Endometrial Hyperplasia (Reproductive system and breast disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No